CLINICAL TRIAL: NCT01663896
Title: Observational Study of Optical Coherence Tomography (OCT) in Patients Undergoing Fractional Flow Reserve (FFR) and Percutaneous Coronary Intervention Stage I (ILUMIEN I)
Brief Title: Observational Study of OCT in a Patients Undergoing FFR
Acronym: ILUMIEN I
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CVD-0612
Record Dates: First submitted 2012-08-07; First posted 2012-08-13 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease
Keywords: OCT, FFR, percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single or multi vessel disease: Pre- and post-PCI fractional flow reserve (FFR) and OCT were performed in participants.
  Interventions: Device: OCT stent guidance

INTERVENTIONS:
Device: OCT stent guidance — Participants undergoing pre- and post-PCI fractional flow reserve (FFR) and OCT

SUMMARY:
The purpose of this study is to define and evaluate optical coherence tomography (OCT) stent guidance parameters through prospective data collection in percutaneous coronary intervention (PCI) procedures of de novo lesions.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) is an imaging modality that uses near-infrared light to produce high resolution, real-time images that are clearer and more quickly produced than those produced by intravascular ultrasound (IVUS). OCT imaging is performed utilizing an imaging catheter with a single optical fiber core that both emits light and records its reflection while simultaneously rotating 360° during continuous pullback within the coronary artery. Fractional Flow Reserve (FFR) is a pressure-derived, lesion-specific, physiological index determining the hemodynamic severity of intracoronary lesions. FFR is measured by placing a pressure guidewire across the lesion of interest and pharmacologically inducing hyperemia. The ratio of distal to proximal pressure allows the physician to physiologically determine if the narrowing is the cause of ischemia. the goal of this study is to define new parameters for stent optimization, benefitting from the unique Fourier-domain (FD-OCT) capabilities.

This stage I study will identify the parameters which will be prospectively tested in a second stage II protocol.

In hospital, 30 day, and 12 month outcomes data will be correlated with OCT baseline findings in order to identify optimal stent implant parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient provides signed written informed consent before any study-specific procedure.
3. De novo coronary artery disease in target vessel.
4. Single or multi vessel disease. For multi vessel disease up to two vessels and three lesions treated, with no more than two lesions per vessel. Vessel is defined as, left anterior descending, left circumflex, and right coronary arteries. Any branch within the vessel is considered part of the vessel.
5. Elective or ad hoc PCI, stable angina, acute coronary syndrome (unstable angina and NSTEMI).
6. Angiographically significant (>50% visual estimation) stenosis present in at least one native coronary artery.
7. Mandatory use of FFR and OCT pre and post PCI. PCI strongly recommended in subjects with an FFR ≤ 0.80 in target vessel.

Exclusion Criteria:

1. Subjects with STEMI, emergent PCI, or in cardiogenic shock.
2. Subjects with target left main lesion.
3. Subjects with restenosis or stent thrombosis in the target vessel.
4. Planned use of bare metal stent.
5. Known renal insufficiency (examples being but not limited to eGFR < 60 ml/kg/m2, serum creatinine ≥ 2.5 mg/dL, or on dialysis).
6. Aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
7. Extreme angulation (> 90°) or excessive tortuosity (> two 45° angles) proximal to or within the target lesion.
8. Vessel(s) and lesion(s) not amenable for PCI, for example diffuse disease.
9. Any other medical condition that in the opinion of the investigator will interfere with patient safety or study results.
10. Currently participating in another clinical study that interferes with study results.
11. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure.
12. Life expectancy less than 1 year.
13. Potential for non-compliance to protocol requirements and follow-up.
14. Planned or prior heart transplantation or listed for heart transplant.
15. Any condition that precludes the subject from undergoing PCI, for example subjects with heparin induced thrombocytopenia, or contrast allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective or ad hoc PCI, stable angina, acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2015-03-12 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (15):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Scripps Clinic, Green Hospital, La Jolla, California
  - Florida Hospital Orlando, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Chicago, Maywood, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Baptist Health East, Louisville, Kentucky
  - St. Luke's Hospital/Mid America Heart, Kansas City, Missouri
  - Rutgers Cardiovascular Institute, New Brunswick, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Heart Hospital of Austin, Austin, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- The Prince Charles Hospital, Chermside, Queensland, Australia
- Med. Univ. Vienna, Vienna, Austria
- Belgium (2):
  - OLV Hospital, Aalst
  - Gasthuisberg Leuven, Leuven
- Montreal Heart Institute, Montreal, Quebec, Canada
- University of Hong Kong, Hong Kong, Hong Kong, China
- University Hospital Brno, Brno, Czechia
- France (3):
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHC du Marie Lannelongue, Le Plessis-Robinson
  - Clinique Pasteur, Toulouse
- Deutsches Herzzentrum, Munich, Germany
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Centro Cardiologico Monzino, Milan
  - Ospedale San Giovanni Addolorata, Rome
- Japan (4):
  - Kobe University Graduate School of Medicine, Hyōgo
  - Nara Medical University Hospital, Nara
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Wakayama Medical University, Wakayama
- Thoraxcentre Erasmus MC, Rotterdam, Netherlands
- Hospital Univ. Clinico San Carlos, Madrid, Spain
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijns W, Shite J, Jones MR, Lee SW, Price MJ, Fabbiocchi F, Barbato E, Akasaka T, Bezerra H, Holmes D. Optical coherence tomography imaging during percutaneous coronary intervention impacts physician decision-making: ILUMIEN I study. Eur Heart J. 2015 Dec 14;36(47):3346-55. doi: 10.1093/eurheartj/ehv367. Epub 2015 Aug 4. PMID 26242713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially a total of 1069 subjects gave consent from 36 investigational sites, of which 418 qualified subjects completed enrollment in February 2014 at 35 investigational sites. First subject was enrolled on Dec 11, 2012 and the last subject completed the 12 month follow-up on Mar 12, 2015.
Pre-assignment Details: Of the 1069 subjects, 616 were failed to screen and 35 were not qualified for inclusion. Thus 418 subjects underwent pre-intervention fractional flow reserve (FFR) and optical coherence tomography (OCT), percutaneous coronary intervention (PCI), and post intervention FFR and OCT. The subjects were followed up through 12 month post stent implant.
Groups:
- Optical Coherence Tomography (OCT): Participants undergoing PCI with intention to perform FFR and OCT pre and post PCI.
Period: Overall Study
Arm/Group | Optical Coherence Tomography (OCT)
Started | 418
Completed | 375
Not Completed | 43
Not completed — Various reasons | 43

BASELINE CHARACTERISTICS:
Arm/Group | Optical Coherence Tomography (OCT)
Number analyzed (Participants) | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 314
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 153
  Czechia | 14
  Japan | 97
  United Kingdom | 7
  Spain | 11
  Canada | 4
  Austria | 5
  Netherlands | 4
  Belgium | 44
  China | 25
  Italy | 32
  Australia | 11
  France | 5
  Germany | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of OCT Peri-procedural Guidance Parameter(s) for Stenting
Description: Incidence of OCT peri-procedural guidance parameter(s) for stenting and their relation to patient outcomes in-hospital.
Time Frame: In-hospital until discharge
Measure: Number; unit: Percentage of per-subject incidence
Groups:
- Optical Coherence Tomography (OCT): A subject who provides a signed Informed Consent Form, meets eligibility criteria, undergoes angiography and pre-intervention FFR, OCT, PCI, and post intervention FFR and OCT.
Arm/Group | Optical Coherence Tomography (OCT)
Number analyzed (Participants) | 418
Percentage of per-subject incidence
  Device-oriented MACE (Cardiac death) | 0
  Device-oriented MACE(MI-AEC definition) | 6.7
  Device-oriented MACE(MI-3rd Universal definition) | 6.2
  Device-oriented MACE(TLR) | 0.2
  Patient-oriented MACE(All-cause mortality) | 0.2
  Patient-oriented MACE(MI-ARC Definition) | 6.7
  Patient-oriented MACE(MI-3rd Universal definition) | 6.2
  Patient-oriented MACE(Any Revascularization) | 0.2
  Stent Thrombosis(Definite) | 0
  Stent Thrombosis(Probable) | 0
  Stent Thrombosis(Possible) | 0
  Stent Thrombosis(Early) | 0
  Stent Thrombosis(Late) | 0
  Stent Thrombosis(Very Late) | 0

2. Primary Outcome: Incidence of OCT Peri-procedural Guidance Parameter(s) for Stenting
Description: Incidence of OCT peri-procedural guidance parameter(s) for stenting and their relation to patient outcomes through 30 days
Time Frame: 30 Days
Measure: Number; unit: Percentage of per-subject incidence
Arm/Group | Optical Coherence Tomography (OCT)
Number analyzed (Participants) | 416
Percentage of per-subject incidence
  Device-oriented MACE (Cardiac death) | 0
  Device-oriented MACE(MI-AEC definition) | 7.2
  Device-oriented MACE(MI-3rd Universal definition) | 6.7
  Device-oriented MACE(TLR) | 0.7
  Patient-oriented MACE(All-cause mortality) | 0.2
  Patient-oriented MACE(MI-ARC Definition) | 7.9
  Patient-oriented MACE(MI-3rd Universal definition) | 7.5
  Patient-oriented MACE(Any Revascularization) | 1.7
  Stent Thrombosis(Definite) | 0
  Stent Thrombosis(Probable) | 0
  Stent Thrombosis(Possible) | 0
  Stent Thrombosis(Early) | 0.2
  Stent Thrombosis(Late) | 0
  Stent Thrombosis(Very Late) | 0

3. Primary Outcome: Incidence of OCT Peri-procedural Guidance Parameter(s) for Stenting (Academic Research Consortium(ARC))
Description: Incidence of OCT peri-procedural guidance parameter(s) for stenting and their relation to patient outcomes through 12 months
Time Frame: 12 months
Measure: Number; unit: Percentage of per-subject incidence
Arm/Group | Optical Coherence Tomography (OCT)
Number analyzed (Participants) | 399
Percentage of per-subject incidence
  Device-oriented MACE (Cardiac death) | 0
  Device-oriented MACE(MI-AEC definition) | 8.3
  Device-oriented MACE(MI-3rd Universal definition) | 7.8
  Device-oriented MACE(TLR) | 2.5
  Patient-oriented MACE(All-cause mortality) | 1.8
  Patient-oriented MACE(MI-ARC Definition) | 9.3
  Patient-oriented MACE(MI-3rd Universal definition) | 8.8
  Patient-oriented MACE(Any Revascularization) | 5.5
  Stent Thrombosis(Definite) | 0.3
  Stent Thrombosis(Probable) | 0
  Stent Thrombosis(Possible) | 0.5
  Stent Thrombosis(Early) | 0.3
  Stent Thrombosis(Late) | 0.5
  Stent Thrombosis(Very Late) | 0

4. Secondary Outcome: Percentage of Change in Physician Decision-making Pre and Post PCI Due to OCT
Description: Assessment of OCT on Physician Decision Making includes:
  * Frequency of changes in treatment strategy based on OCT parameter real time assessment vs. angiographic assessment
  * OCT parameters as assessed by Core Lab
Time Frame: 1 Year
Measure: Number; unit: Percentage of participants
Arm/Group | Optical Coherence Tomography (OCT)
Number analyzed (Participants) | 418
Percentage of participants
  Procedure Planning(Pre-PCI OCT) | 57
  Procedure Planning(Post-PCI OCT) | 27
  Physician decision-making (Pre-PCI OCT) | 65
  Physician decision-making (Post-PCI OCT) | 65

ADVERSE EVENTS:
Time Frame: 1-Year
Arm/Group | Optical Coherence Tomography (OCT)
All-Cause Mortality (participants affected / at risk) | 8/418
Serious Adverse Events (participants affected / at risk) | 112/418
Other Adverse Events (participants affected / at risk) | 128/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optical Coherence Tomography (OCT) (N=418)
Abdominal Pain (Gastrointestinal disorders) | 1
Abnormal Lab Value (Investigations) | 2
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute Erosive Gastritis (Gastrointestinal disorders) | 1
Anemias (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Arterial Hypertension/Hypertension (Vascular disorders) | 2
Ascites (General disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 3
Atrial Flutter (Cardiac disorders) | 1
Atrioventricular (AV) Dissociation (Cardiac disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 2
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cardiac Arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiovascular Deconditioning (Cardiac disorders) | 1
Chest Pain (General disorders) | 24
Cholelithiasis (Hepatobiliary disorders) | 1
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Coronary Artery Disease (Cardiac disorders) | 2
Diabetic Ketoacidosis (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Discomfort (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
EKG Abnormalities (Investigations) | 1
Echo Finding (Investigations) | 1
Elective Surgery (Surgical and medical procedures) | 1
Emesis/Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 6
Gingival Bleeding (General disorders) | 1
Gout (Musculoskeletal and connective tissue disorders) | 1
Heart Failure (Cardiac disorders) | 2
Hematochezia (General disorders) | 1
Hematoma (Vascular disorders) | 5
Hematuria (Renal and urinary disorders) | 1
Hyperkalemia (Investigations) | 1
Hypotension (Vascular disorders) | 2
Idiopathic Interstitial Lung Diseases (Respiratory, thoracic and mediastinal disorders) | 1
Influenza (Infections and infestations) | 1
Intracerebral Haemorrhage (Nervous system disorders) | 1
Ischemic Stroke (Nervous system disorders) | 1
Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Left Bundle Branch Block/Complete Left Bundle Branch Block (Cardiac disorders) | 1
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melena (General disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myocardial Infarction (Cardiac disorders) | 8
Non-Cardiac Chest Pain (General disorders) | 1
Non-Endpoint Transient Ischemic Attack (TIA) (Nervous system disorders) | 1
Other (General disorders) | 14
Pericardial Tamponade (Cardiac disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia in the Compromised Host (Infections and infestations) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Side Branch Compromise (Injury, poisoning and procedural complications) | 1
Stroke (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 1
Unstable Angina (Cardiac disorders) | 3
VASC Vessel Stenosis (Vascular disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 2
Vessel Stenosis (Vascular disorders) | 10
Visual Disturbance (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optical Coherence Tomography (OCT) (N=418)
Abdominal Pain (General disorders) | 1
Abnormal Lab Value (Investigations) | 1
Abrasion (General disorders) | 1
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Acute Pancreatitis (Gastrointestinal disorders) | 1
Allergy (Immune system disorders) | 1
Anemias (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Anxiety (Psychiatric disorders) | 1
Aortic Aneurysms (Vascular disorders) | 1
Apnea (General disorders) | 1
Arm Fracture (Musculoskeletal and connective tissue disorders) | 2
Arm Pain (Musculoskeletal and connective tissue disorders) | 1
Arterial Hypertension/Hypertension (Vascular disorders) | 5
Arteriovenous (AV) Fistula (Vascular disorders) | 1
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Infections and infestations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Back Pain (General disorders) | 1
Bleeding (Vascular disorders) | 2
Blurred Vision (Eye disorders) | 1
Bruise/Purpura Simplex (Skin and subcutaneous tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Callus (General disorders) | 1
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal Tunnel (Nervous system disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Chest Pain (General disorders) | 18
Chest Tightness (General disorders) | 4
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 4
Chronic Renal Failure (Renal and urinary disorders) | 1
Common Cold/Upper Respiratory Tract Infection (Infections and infestations) | 6
Conjunctivitis (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Difficulty Catching Breath (Respiratory, thoracic and mediastinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Dizziness (Ear and labyrinth disorders) | 5
Dry Eyes (Eye disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Dysuria (Renal and urinary disorders) | 1
EKG Abnormalities (Investigations) | 4
Edema (General disorders) | 3
Eye Infection (Eye disorders) | 1
Fainting/Blackout (Nervous system disorders) | 1
Fatigue/Generalized Fatigue (General disorders) | 10
Fever (Infections and infestations) | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gout (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 4
Hiatus Hernia (Gastrointestinal disorders) | 1
Hip Pain (General disorders) | 5
Hyperglycemia (Endocrine disorders) | 2
Hypokalemia (Investigations) | 1
Hypokinetic Septal Motion (Cardiac disorders) | 1
Hyponatremia (Investigations) | 1
Ingestion (Gastrointestinal disorders) | 1
Iron-Deficiency Anemia (Blood and lymphatic system disorders) | 1
Knee Pain (General disorders) | 5
Lacerations (General disorders) | 1
Low Back Pain (Musculoskeletal and connective tissue disorders) | 4
Melena (General disorders) | 1
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 1
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5
Myalgias (General disorders) | 1
Nausea (General disorders) | 1
Neck Pain (General disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Obstructive Sleep Apnea (General disorders) | 2
Orthostatic Hypotension (Vascular disorders) | 1
Other (General disorders) | 14
Pain (General disorders) | 5
Palpitations (Cardiac disorders) | 2
Peak T Waves (Investigations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Post-Nasal Drainage (General disorders) | 1
Premature Ventricular Contraction (Cardiac disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Renal Artery Stenosis (Vascular disorders) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin Bruise (Skin and subcutaneous tissue disorders) | 1
Skin Lesions (Skin and subcutaneous tissue disorders) | 2
Swelling (General disorders) | 1
Syncope (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Thrombus (Vascular disorders) | 1
Tooth Infection (General disorders) | 1
Toothache (General disorders) | 1
Trauma (Injury, poisoning and procedural complications) | 1
Unsustained/Nonsustained Ventricular Tachy/Cardiac Arrhythmia (Cardiac disorders) | 1 — Unsustained/Nonsustained Ventricular Tachy/Cardiac Arrhythmia includes: Other - Non-sustained runs of VT, Ventricular Ectopic Beats/Premature Ventricular Contractions/Premature Ventricular Beats
Urinary Tract Infections (Renal and urinary disorders) | 4
VASC Bruise (Vascular disorders) | 1
VASC Hematoma (Vascular disorders) | 1
VASC Pseudoaneurysm (Vascular disorders) | 1
VASC Vessel Stenosis (Vascular disorders) | 1
Vaso Vagal Response (Nervous system disorders) | 1
Vertigo (Nervous system disorders) | 1
Vessel Stenosis (Vascular disorders) | 3
Viral Gastroenteritis (Gastrointestinal disorders) | 1
Visual Disturbance (Eye disorders) | 2
Weakness (General disorders) | 1
Wrist Sprain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Patients with acute STEMI, left main PCI, severe chronic kidney disease, and other high-risk features were excluded. No prescriptive recommendations were provided in the protocol, a wide variation in physician behavior was expected and observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposals for all publications, abstracts, presentations, or journal manuscripts arising from, or related to the Study will be submitted for approval to the Publications Committee. Accordingly, decisions on timing and content of publications and presentations from the Study will be coordinated with the Study Publication Committee and Sponsor.